CLINICAL TRIAL: NCT05095493
Title: Oral Zinc Supplementation to Enhance Effects of Botulinum Neurotoxin Injection: an n of 1 Study
Brief Title: Oral Zinc Supplementation to Enhance Botulinum Neurotoxin Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Padraig O'Suilleabhain, Professor of Neurology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-082021-075
Record Dates: First submitted 2021-10-01; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Dystonia, Focal
MeSH Terms: conditions — Dystonic Disorders | interventions — Zinc Acetate

STUDY DESIGN:
Intervention Model Description: Single site randomized placebo controlled trial, cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy prepares vials labeled A and B, and reveals code to PI after data lock
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zinc, then placebo (Experimental): Participants first received oral zinc acetate 50 mg tab each day for 7 days before scheduled BoNT injection. 3 months later participants received oral placebo (matching oral zinc) tablet each day for 7 days before scheduled BoNT injection.
  Interventions: Dietary Supplement: Zinc Acetate; Dietary Supplement: Placebo
- placebo, then zinc (Experimental): Participants first received placebo tablet (matching oral zinc) each day for 7 days before scheduled BoNT injection. 3 months later participants received oral zinc acetate 50 mg tablet each day for 7 days before scheduled BoNT injection.
  Interventions: Dietary Supplement: Zinc Acetate; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc Acetate — 50 mg tablet
Dietary Supplement: Placebo — Zinc Acetate matched placebo tablet

SUMMARY:
Botulinum neurotoxin (BoNT) is injected into muscles for treatment of dystonia. BoNTs are zinc proteases, and their enzymatic effect is reduced in the setting of low zinc. The study hypothesis is that a large enough fraction of unselected dystonia patients receiving BoNT injection have suboptimal zinc concentration in their tissues, and will experience improved response to BoNT if the injection is preceded by oral zinc supplementation (OZS). OZS consists of 50 mg of zinc acetate oral tablet each day for 7 days before injection. This is a double blind placebo controlled cross-over study, randomized order placebo and OZS, in patients at a neurology clinic on stable dose of BoNT.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the PI
* Age 18-80
* Male or female
* With an approved indication for BoNT such as dystonia or hemifacial spasm
* Have received either two or three BoNT injection cycles within the prior 8 months
* Prior two injection cycles length differed by no more than 2 weeks
* Prior two injection cycles used same brand of BoNT and similar dose within 15%

Exclusion Criteria:

* Concommitant use of penicillamine or cisplatin

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change | End of study, week 48
  Patient selects one of three options: My response to BoNT injection with bottle A tablets was overall better than with bottle B tablets; My response to BoNT injection with bottle B tablets was overall better than bottle A tablets; or Neither BoNT injection with bottle A or with bottle B tablets was overall better than the other

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | At study visits 3 and 4, which are 3 months after the BoNT injection cycles with intervention OZS or placebo
  Unstructured interview soliciting side-effects in the interval since prior BoNT injection

CONTACTS AND LOCATIONS:
Overall Officials: Padraig E O'Suilleabhain, MD, Principal Investigator — UTSW

IPD SHARING:
Plan to Share IPD: No